CLINICAL TRIAL: NCT00651326
Title: A Phase III Study of Neoadjuvant Docetaxel and Androgen Suppression Plus Radiation Therapy Versus Androgen Suppression Alone Plus Radiation Therapy for High-Risk Localized Adenocarcinoma of the Prostate
Brief Title: Androgen Suppression and Radiation With/Out Docetaxel in High-Risk Localized Prostate Cancer
Acronym: DART
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PR12; CAN-NCIC-PR12 (Registry Identifier: PDQ); CDR0000589247 (Other: PDQ)
Record Dates: First submitted 2008-04-01; First posted 2008-04-02 (Estimated); Last update posted 2023-08-04 (Actual); Status verified 2020-03

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage I prostate cancer; stage II prostate cancer; stage III prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — bicalutamide; Buserelin; Flutamide; Goserelin; Leuprolide; Neoadjuvant Therapy; Radiotherapy; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antiandrogen; LHRH; Docetaxel, Radiation Therapy (Active Comparator): Antiandrogen (Flutamide or Bicalutamide) LHRH agonist (Eligard) Docetaxel
  Interventions: Drug: bicalutamide; Drug: buserelin; Drug: flutamide; Drug: goserelin; Drug: leuprolide acetate; Procedure: neoadjuvant therapy; Procedure: quality-of-life assessment; Radiation: radiation therapy; Drug: Docetaxel
- Antiandrogen; LHRH; Radiation Therapy (Active Comparator): Antiandrogen (Flutamide or Bicalutamide) LHRH agonist (Eligard)
  Interventions: Drug: bicalutamide; Drug: buserelin; Drug: flutamide; Drug: goserelin; Drug: leuprolide acetate; Procedure: neoadjuvant therapy; Procedure: quality-of-life assessment; Radiation: radiation therapy

INTERVENTIONS:
Drug: bicalutamide
Drug: buserelin
Drug: flutamide
Drug: goserelin
Drug: leuprolide acetate
Procedure: neoadjuvant therapy
Procedure: quality-of-life assessment
Radiation: radiation therapy — 46 Gy in 23 fractions over < 5 weeks.
  Boost:
  24-28 Gy in 12-14 fractions over < 3 weeks
Drug: Docetaxel
  Arms: Antiandrogen; LHRH; Docetaxel, Radiation Therapy

SUMMARY:
RATIONALE: Androgens can cause the growth of prostate cancer cells. Antihormone therapy, such as flutamide, bicalutamide, leuprolide, buserelin, and goserelin, may lessen the amount of androgens made by the body. Radiation therapy uses high-energy x-rays to kill tumor cells. Drugs used in chemotherapy, such as docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. It is not yet known whether giving androgen suppression therapy together with radiation therapy is more effective with or without docetaxel in treating prostate cancer.

PURPOSE: This randomized phase III trial is studying androgen suppression therapy, radiation therapy, and docetaxel to see how well they work compared with androgen suppression therapy and radiation therapy in treating patients with high-risk localized prostate cancer.

CLOSURE: This trial closed to further accrual in November 2009. The study endpoints will not be reached.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To compare disease-free survival rates in patients with high-risk localized adenocarcinoma of the prostate treated with androgen suppression therapy and radiotherapy with vs without docetaxel.

Secondary

* To compare overall survival.
* To compare time to biochemical disease progression.
* To compare time to local disease progression.
* To compare time to distant disease progression.
* To compare time to next anticancer therapy.
* To compare progression-free survival.
* To compare degree of prostate-specific antigen (PSA) suppression prior to radiotherapy.
* To compare quality of life (QOL) using EORTC QLQ C30 and EORTC QLQ PR25 questionnaires and a trial-specific checklist.
* To compare the nature, severity, and frequency of adverse events.

OUTLINE: This is a multicenter study. Patients are stratified according to Gleason score (≤ 7 vs ≥ 8), baseline prostate-specific antigen (PSA) (> 20 ng/mL vs ≤ 20 ng/mL), and participating center. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive androgen suppression therapy comprising oral flutamide three times daily or oral bicalutamide once daily for 4 weeks AND leuprolide subcutaneously (SC) or intramuscularly every 1-6 months, buserelin SC every 2 or 3 months, or goserelin SC every 1 or 3 months for 3 years. Patients also receive docetaxel IV over 60 minutes on day 1. Treatment with docetaxel repeats every 21 days for up to 4 courses. Beginning at least 4 weeks after completion of chemotherapy, patients undergo pelvic radiotherapy once daily 5 days a week for up to 8 weeks.
* Arm II: Patients receive androgen suppression therapy and undergo pelvic radiotherapy as in arm I.

Patients complete quality of life questionnaires at baseline, periodically during treatment, and then every 6 months for 5 years.

After completion of study treatment, patients are followed at 3 and 6 months, every 6 months for 5 years, and then annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate

  * Localized (N0, M0) disease
  * No small cell or transitional cell carcinoma in the biopsy specimen
* Considered to be at high risk for recurrence based on the presence of at least one of the following adverse prognostic features:

  * T stage ≥ 3a
  * Gleason score ≥ 8
  * Baseline prostate-specific antigen (PSA) > 20 ng/mL
* Deemed to be an appropriate candidate for chemotherapy, as assessed by a medical oncologist
* Negative pelvic and para-aortic lymph nodes on CT scan or MRI of the abdomen and pelvis

  * Any lymph node appearing ≥ 1.5 cm on CT scan or MRI must be histologically negative by either needle aspirate or lymph node dissection
* No metastases by chest x-ray and bone scan

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 10.0 g/dL
* AST and/or ALT ≤ 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 2.5 times ULN
* Total bilirubin normal
* Serum creatinine ≤ 1.5 times ULN
* Able (i.e., sufficiently fluent) and willing to complete the quality of life questionnaires in either English or French
* Fertile patients must use effective contraception
* No history of other malignancies, except adequately treated nonmelanoma skin cancer or other curatively treated solid tumor with no evidence of disease for > 5 years
* No serious non-malignant disease resulting in a life expectancy of < 10 years
* No known hypersensitivity to any study medications
* No existing peripheral neuropathy ≥ grade 2
* No bilateral hip replacement prostheses
* No contraindication to pelvic radiotherapy including, but not limited to, inflammatory bowel disease or severe bladder irritability
* No medical condition that would contraindicate the study treatment regimen, including severe respiratory insufficiency, uncontrolled diabetes, or severe hypertension
* No other serious illness or psychiatric or medical condition that would preclude management of the patient according to the study, including active uncontrolled infection or significant cardiac dysfunction

PRIOR CONCURRENT THERAPY:

* Prior androgen suppression therapy allowed provided it was initiated no more than 4 weeks prior to study entry
* At least 4 weeks since prior 5-alpha-reductase inhibitors (e.g., finasteride) for benign prostatic hypertrophy
* No prior cytotoxic anticancer therapy
* No prior chemotherapy for carcinoma of the prostate
* No prior surgical treatment for carcinoma of the prostate, except transurethral resection or bilateral orchiectomy
* No prior pelvic radiotherapy
* No concurrent nilutamide
* No other concurrent investigational drugs
* No other concurrent anticancer therapy (cytotoxic therapy, biologic/immunotherapy, or radiotherapy)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2008-06-02 (Actual); Primary Completion 2010-05-14 (Actual); Study Completion 2011-01-18 (Actual)

PRIMARY OUTCOMES:
Disease-free survival

SECONDARY OUTCOMES:
Overall survival
Time to biochemical disease progression
Time to local disease progression
Time to distant disease progression
Time to next anti-cancer therapy
Progression-free survival
Degree of prostate-specific antigen (PSA) suppression prior to radiotherapy
Quality of life
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Michael R. McKenzie, MD, FRCPC, Study Chair — British Columbia Cancer Agency; Kim N. Chi, MD, Study Chair — British Columbia Cancer Agency
Locations (13):
- Canada (13):
  - Tom Baker Cancer Centre, Calgary
  - Cross Cancer Institute, Edmonton
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton
  - BCCA - Cancer Centre for the Southern Interior, Kelowna
  - London Regional Cancer Program, London
  - Credit Valley Hospital, Mississauga
  - McGill University - Dept. Oncology, Montreal
  - Lakeridge Health Oshawa, Oshawa
  - Ottawa Health Research Institute - General Division, Ottawa
  - Saskatoon Cancer Centre, Saskatoon
  - Univ. Health Network-Princess Margaret Hospital, Toronto
  - BCCA - Vancouver Cancer Centre, Vancouver
  - CancerCare Manitoba, Winnipeg

IPD SHARING:
Plan to Share IPD: No